CLINICAL TRIAL: NCT01761526
Title: Parallel Group Trial to Evaluate the Pharmacokinetics and Safety / Tolerability of Single-Dose Treatment With Rotigotine Continuous Delivery System (10 cm2 / 4.5 mg) in Japanese and Caucasian Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetics (PK), Safety, Tolerability of Single-Dose Transdermal Rotigotine in Japanese and Caucasian Healthy Male / Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: Schwarz BioSciences GmbH (Unknown); Alfred-Nobel-Str. 10 (Unknown); 40789 Monheim am Rhein (Unknown)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SP0717
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Rotigotine; Neupro; Japanese; Caucasian; Male; Female; Single dose; Pharmacokinetics
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine in Healthy Japanese (Experimental): * Rotigotine transdermal patch
  * Single dose application of 2 mg / 24 hours Rotigotine in Healthy Japanese subjects
  * Transdermal patch over 24 hours
  Interventions: Drug: Rotigotine transdermal patch
- Rotigotine in Caucasian (Experimental): * Rotigotine transdermal patch
  * Single-Dose application of 2 mg / 24 hours Rotigotine in healthy Caucasian subjects
  * Transdermal patch over 24 hours
  Interventions: Drug: Rotigotine transdermal patch

INTERVENTIONS:
Drug: Rotigotine transdermal patch — Rotigotine transdermal patch, single-dose application over 24 hours 2 mg /24 hours (10 cm2)
  Other Names: Neupro

SUMMARY:
To investigate the Pharmacokinetics (PK) of transdermally delivered Rotigotine in Japanese and Caucasian Female and Male Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy according to assessments done at eligibility assessment (medical history, physical examination, blood pressure, heart rate, Electrocardiogram (ECG), hematology, clinical chemistry, urinalysis)
* Subject is of normal body-weight as determined by a body mass index ranging between 18 to 28 kg / m²
* Subject is Japanese or Caucasian. Japanese subjects are born in Japan and left Japan not more than 10 years ago. Both parents of the Japanese subjects are 100 % Japanese

Exclusion Criteria:

* Subjects (females) without medically adequate contraception (e.g. mechanical contraception (Intrauterine-Device IUD), sterilization, hysterectomy) or on lactation or pregnant women. Subjects with oral contraception or hormone replacement within 4 weeks prior to eligibility assessment
* Subject has a history of chronic alcohol or drug abuse
* Subject has a consumption of more than 20 g of alcohol / day (amount corresponds to 0.5 l of beer / day or 0.25 l of wine / day or 3 glasses (à 2 cl) of liquor / day
* Subject has a clinically relevant allergy
* Subject has a known or suspected drug hypersensitivity in particular, to any component of the trial medication
* Subject has any clinically significant abnormality in physical examination
* Subject has a heart rate at rest less than 50 beats per minute (bpm) or more than 100 bpm
* Subject has systolic blood pressure lower than 100 mmHg or higher than 145 mmHg or diastolic blood pressure higher than 95 mmHg or lower than 60 mmHg
* Subject has an atopic or eczematous dermatitis and / or an active skin disease or skin tumors
* Subject has a history of significant skin hypersensitivity to adhesives or other transdermal products or recent unresolved contact dermatitis

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2002-10; Primary Completion 2002-10 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) from zero up to the last measured concentration greater than the Lower Limit of Quantitation (LOQ) [AUC (0-t)] of unconjugated Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero up to the last measured concentration greater than the Lower Limit of Quantitation (LOQ) normalized [AUC (0-t)norm] of unconjugated Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Maximum concentration in plasma [Cmax] of unconjugated Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Maximum concentration in plasma normalized by body weight [Cmax,norm] of unconjugated Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero up to the last measured concentration greater than the Lower Limit of Quantitation (LOQ) [AUC (0-t)] of total Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Maximum concentration in plasma [Cmax] of total Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Maximum concentration in plasma normalized by body weight [Cmax,norm] of total Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero up to the last measured concentration greater than the Lower Limit of Quantitation (LOQ) [AUC (0-t)] of total Despropylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero up to the last measured concentration greater than the Lower Limit of Quantitation (LOQ) normalized by body weight [AUC (0-t)] of total Despropylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Maximum concentration in plasma [Cmax] of total Despropylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Maximum concentration in plasma normalized by body weight [Cmax,norm] of total Despropylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero up to the last measured concentration greater than the Lower Limit of Quantitation (LOQ) [AUC (0-t)] of total Desthienylethylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero up to the last measured concentration greater than the Lower Limit of Quantitation (LOQ) normalized by body weight [AUC (0-t)] of total Desthienylethylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Maximum concentration in plasma [Cmax] of total Desthienylethylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Maximum concentration in plasma normalized by body weight [Cmax, norm] of total Desthienylethylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose

SECONDARY OUTCOMES:
Terminal half-life [t1/2] of unconjugated Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Time of maximum concentration [tmax] of unconjugated Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero to infinity [AUC (0-inf)] of unconjugated Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Total body clearance (CL) of unconjugated Rotigotine normalized by body weight (BW) [CL/f/BW] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Apparent volume of distribution of unconjugated Rotigotine normalized by body weight [Vz/f/BW] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Amounts of unconjugated Rotigotine excreted in urine [Ae] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Fraction of unconjugated Rotigotine excreted into urine [fe (% of dose)] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Renal Clearance [CLR] of unconjugated Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Terminal half-life [t1/2] of total Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Time of maximum concentration [tmax] of total Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero to infinity [AUC (0-inf)] of total Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Total body clearance of total Rotigotine normalized by body weight [CL/f/BW] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Apparent volume of distribution normalized of total Rotigotine by body weight [Vz/f/BW] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Amount of total Rotigotine excreted into urine [Ae] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Fraction of total Rotigotine excreted into urine [fe (% of dose)] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Renal clearance [CLR] of total Rotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Terminal half-life [t1/2] of total Despropylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Time of maximum concentration [tmax] of total Despropylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero to infinity [AUC (0-inf)] of total Despropylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Total body clearance of total Despropylrotigotine normalized by body weight [CL/f/BW] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Apparent volume of distribution of total Despropylrotigotine normalized by body weight [Vz/f/BW] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Amount of total Despropylrotigotine excreted into urine [Ae] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Fraction of total Despropylrotigotine excreted into urine [fe (% of dose)] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Renal Clearance [CLR] of total Despropylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Terminal half-life [t1/2] of total Desthienylethylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Time of maximum concentration [tmax] of total Desthienylethylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Area under the concentration-time curve from zero to infinity [AUC (0-inf)] of total Desthienylethylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Total body clearance of total Desthienylethylrotigotine normalized by body weight [CL/f/BW] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Apparent volume of distribution of total Desthienylethylrotigotine normalized by body weight [Vz/f/BW] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Amount of total Desthienylethylrotigotine excreted into urine [Ae] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Fraction of total Desthienylethylrotigotine excreted into urine [fe (%of dose)] | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose
Renal clearance [CLR] of total Desthienylethylrotigotine | From Baseline (0 hours Pre-Dose) up to 60 hours Post-Dose
  Blood sampling at 0 hours (Pre-Dose), 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 25 hours, 26 hours, 28 hours, 30 hours, 33 hours, 36 hours, 48 hours, and 60 hours Post-Dose

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 01, Neuss, Germany